CLINICAL TRIAL: NCT04714762
Title: eHealth in Treatment of Gestational Diabetes - eMOM GDM -Study (Phase 2)
Brief Title: eHealth in Treatment of Gestational Diabetes (eMOMGDM)
Acronym: eMOMGDM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other); Aalto University (Other); UKK Institute (Other); Tampere University (Other); Finnish Institute for Health and Welfare (Other Government); Fujitsu (Unknown); Elisa Oyj (Unknown); Business Finland (Other)
Responsible Party: Principal Investigator, Saila Koivusalo, MD Adjunct prof, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUS/2165/2018-Phase 2
Record Dates: First submitted 2021-01-11; First posted 2021-01-19 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Gestational Diabetes; Mobile Application
Keywords: gestational diabetes; continuous glucose monitoring; physical activity; nutrition; behaviour change; stress; recovery; human-computer interaction; mobile application; self tracking
MeSH Terms: conditions — Diabetes, Gestational; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data will be anonomized (ID coded)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (eMOM GDM application) (Experimental): Participants in the intervention group will use the eMOM GDM -application one week/month. The participants will also receive regular antenatal care in maternity clinics and hospitals. In addition they will meet a study nurse three times during study period (at GW 24-28, at GW 35-37 and 3 mo postpartum).
  Interventions: Device: eMOM GDM application
- Control (No Intervention): Participants in the control group will meet a study nurse 3 times during study period (at GW 24-28, at GW 35-37 and 3 mo postpartum). They also receive regular antenatal care in maternity clinics and hospitals.

INTERVENTIONS:
Device: eMOM GDM application — Participants in the intervention group will use the eMOM GDM -application one week/month.
  eMOM GDM application includes:
  * continuous glucose monitor (CGM, Medtronic)
  * diet (digital food tracker) (min 3 days during one application week)
  * heartrate, stress and physical activity with the wrist-worn activity tracker (Vivosmart 3)
  * weight measured once a week
  The sensors can be worn and the application used during the whole pregnancy (if a mother is interested in)
  Arms: Intervention (eMOM GDM application)

SUMMARY:
The overall aim of the eMOM GDM-project is to develop and evaluate a novel system to clinical decision making and patient behavior change in treatment of GDM, combining diet, physical activity, sleep, heart rate (e.g. stress), and glucose monitoring within a single system (the eMOM GDM application), and linking the developed application tool for the normal health care system in a new way.

In this second phase of the project, the effect of eMOM GDM application on maternal and neonatal outcomes will be evaluated in a randomized controlled study design. The follow-up study continues until 3 months postpartum.

DETAILED DESCRIPTION:
200 women with gestational diabetes will be randomized into the intervention and the control group at gestational week (GW) 24-28.

Participants in the intervention group will use the eMOM GDM -application one week/month until delivery.

The participants in the intervention and the control group visit study nurse 3 times in study period (at GW 24-28 and GW 35-37 and 3 months postpartum).

Both groups also receive regular antenatal care in maternity clinics and hospitals.

Maternal measurements at enrollment, and at 35-37 GW (both groups):

* Laboratory tests: fp-gluc, HbA1c, fp-insu, lipids, hs-CRP
* Fingertips glucose values from glucose meter (belong to normal antenatal care)
* Fasting blood samples for future analyses
* Weight, height, blood pressure (from the antenatal registry and study visits)
* Questionnaires: background (only at enrollment), diet (food frequency questionnaire), depression (EPDS), motivation (TSRQ+PCS), quality of life (15D)
* Physical activity and sedentary behavior with the hip-worn triaxial accelerometer (UKK RM 42)
* Physical activity and heart rate with Firstbeat Bodyguard

Measurements at Birth:

* Cord blood sample
* Placental weight
* Offspring birthweight, height, body composition (PEA POD Cosmed®)

Maternal measurements at 3 months postpartum:

* Laboratory tests: fp-gluc, HbA1c, fp-insu, lipids, hs-CRP
* fp-gluc, 2h postprandial value, as measured during oral glucose tolerance test (OGTT)
* Fasting blood samples for future analyses
* Firstbeat Bodyguard 2 measurement (3 days)
* Depression questionnaire (EPDS)
* Diet questionnaire (FFQ)

Protocol only for the intervention group

- eMOM GDM application: use: 1 application week + 3 normal care weeks repeatedly until delivery

The application includes:

1. continuous glucose monitor (CGM)

   * fingertips glucose calibration according to CGM protocol (twice per day with Medtronic)
2. diet (digital food tracker)

   * 3 days during one application week
   * For ensuring the quality of food record a researcher will phone interview the participant based on her recordings. This is done after each recording period.
3. heartrate, stress and physical activity with the wrist-worn activity tracker (Vivosmart 3)
4. weight measured once a week

Data from the sensors

* Data from users' input to the application
* Technology acceptance questionnaire (UTAUT) after every application week
* Usability questionnaire, after four weeks usage of the eMOM GDM application
* Semi-structured interview

ELIGIBILITY:
Inclusion Criteria:

* GDM diagnoses at 24-28 gestational weeks

Exclusion Criteria:

* type 1 or type 2 diabetes
* use of medication that influences glucose metabolism (such as continuous therapy with oral corticosteroids or metformin)
* multiple pregnancy
* physical disability
* current substance abuse
* severe psychiatric disorder (that complicates participation to the study)
* significant difficulty in cooperating (e.g. inadequate Finnish language skills)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only women have GDM
Enrollment: 200 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in fasting glucose | from gestational weeks 24-28 to gestational weeks 35-37
  change in fasting glucose measured by Huslab (laboratory measurement)

SECONDARY OUTCOMES:
Fingertips fasting glucose values | from gestational weeks 24-28 up to delivery
  Measured with Contour Next One
Fingertips postbrandial glucose values | from gestational weeks 24-28 up to delivery
  Measured with Contour Next One
Fingertips area under the glucose curve | from gestational weeks 24-28 up to delivery
  Measured with Contour Next One
Gestational weight | weight measured at gestational weeks 24-28 and at 35-37 and collected from antenatal card during whole pregnancy and up to delivery
  Measured with Seca Mod 8787041649 (scale) and registered from antenatal card
Postpartum weight | weight measured at 3 months postpartum
  Measured with Seca Mod 8787041649 (scale)
Physical activity level | at gestational weeks 24-28, 35-37 and at 3 months postpartum
  Measured with the accelerometers UKK RM42 and Firstbeat Bodyguard 2
Total diet | at gestational weeks 24-28), 35-37 and at 3 months postpartum
  Measured with a questionnaire (food frequencey questionnaire, FFQ) concerning participant's diet during previous month. FFQ contains questions about the frequency (number of times per day, week, or month) and the amount of foods consumed in units of common serving sizes. Nutritional quality of total diet is assessed based on calculated daily consumption of foods and intake of nutrients. Better nutritional quality is related to e.g. higher intake of fruits and vegetables, wholegrain cereals, fiber and unsaturated fat, and lower intake of added sugar and saturated fat.
Neonatal body fat% | one measure within 0-3 days after birth of the child
  Measured with PEA POD Cosmed
Motivation to manage GDM | at gestational weeks 24-28 and 35-37
  Measured with a motivation questionnaire (TSRQ and PCS). Minimum value is 1 and maximum 5. The higher score means higher autonomous motivation to manage GDM.
Percentage of participants on metformin treatment | up to 42 gestational weeks
  Percentage of participants need for metformin treatment
Percentage of participants on insulin treatment | up to 42 gestational weeks
  Percentage of participants need for insulin treatment
Newborn birthweight and macrosomia | one measure at birth
  Newborn birth weight and macrosomia (birthweight >4kg)
Incidence of neonatal hypoglycemia | within a week from birth
  Percentage of neonatal hypoglycemia requiring intravenous glucose
Incidence of newborn large for gestational age | one measure at birth
  Percentage of newborn with birthweight percentile > + 2 SD
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | gestational weeks 24-28, gestational weeks 35-37, 3 months postpartum
  Change in HOMA-IR measured by Huslab (laboratory measurement), calculated as: fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5.
2-h OGTT | 3 months postpartum
  2-hour blood glucose levels measured with OGTT (75g)
Stress levels | gestational weeks 24-28, gestational weeks 35-37, 3 months postpartum
  Calculated based on dedicated HRV-based algorithm by Firstbeat. Defined as percentages.
Costs | gestational weeks 24-28, 3 months postpartum
  Costs of the intervention and treatment in healthcare. Defined as €/participant.

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Yes
All data will be collected in Helsinki University Hospital Datalake from where pseudo-anonymised data can be requested until 2032 via a data sharing contract. Proposals should be directed to tietopalvelu(a)hus.fi.
Supporting Information: Study Protocol
Time Frame: Until 2032

REFERENCES:
- [Derived] Maattanen S, Koivusalo S, Ylinen H, Heinonen S, Kyto M. The Effect of a Mobile App (eMOM) on Self-Discovery and Psychological Factors in Persons With Gestational Diabetes: Mixed Methods Study. JMIR Mhealth Uhealth. 2025 Jun 4;13:e60855. doi: 10.2196/60855. PMID 40466096
- [Derived] Kyto M, Markussen LT, Marttinen P, Jacucci G, Niinisto S, Virtanen SM, Korhonen TE, Sievanen H, Vaha-Ypya H, Korhonen I, Heinonen S, Koivusalo SB. Comprehensive self-tracking of blood glucose and lifestyle with a mobile application in the management of gestational diabetes: a study protocol for a randomised controlled trial (eMOM GDM study). BMJ Open. 2022 Nov 7;12(11):e066292. doi: 10.1136/bmjopen-2022-066292. PMID 36344008